CLINICAL TRIAL: NCT00472134
Title: Prospective, Randomized, Double-blind Trial of Continuous Infusion of 0.5% Bupivacaine be Elastomeric Pump for Prospective Pain Management After Laparoscopic Ventral Hernia Repair.
Brief Title: Laparoscopic Ventral Hernia Repair With Elastomeric Pain Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Michael J. Rosen, MD., Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 11-05-22
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2012-01

CONDITIONS: Hernia, Ventral
Keywords: Hernia; Ventral; Laparoscopic Hernia Repair
MeSH Terms: conditions — Hernia, Ventral; Hernia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivicaine via Elastomeric pump (Active Comparator): Bupivicaine via elastomeric pump
  Interventions: Drug: bupivacaine
- Placebo via elastomeric pump (Placebo Comparator): Placebo via elastomeric pump
  Interventions: Device: On-Q PainBuster pump

INTERVENTIONS:
Drug: bupivacaine — administered locally, 0.5% Bupivacaine (Marcaine Abbott Laboratories) or saline administered continuously for 48 hours at 2 mL/h.
  Other Names: Marcaine
  Arms: Bupivicaine via Elastomeric pump
Device: On-Q PainBuster pump — local anesthetic (bupivacaine) administered via a pain relief system consisting of a 20 gauge soaker catheter attached to an elastomeric balloon pump that is capable of infusing a set volume of local anesthetic over a wide area of surgical site for 2 to 5 days
  Arms: Placebo via elastomeric pump

SUMMARY:
The purpose of this study is to determine the effects of a local anesthetic dispensed via a tiny catheter device, called the ON-Q PainBuster pump, placed during surgery on top of the mesh used in the laparoscopic repair of ventral hernias. The goals are:

* reducing postoperative pain from this procedure
* decreasing length of hospital stay
* reducing or eliminating amount of post-operative narcotics used

DETAILED DESCRIPTION:
One outcome of the greater than 2 million abdominal operations performed in the United States each year is an incisional hernia rate of 3% to 20%. As a result, approximately 150,000 ventral hernia repairs are performed annually. The increasing number of incisional hernias merely reflects the evolution of surgery with the ability to perform larger abdominal operations such as aortic surgery and colectomy. Primary tissue repairs have had unacceptable rates of recurrence when used for larger defects. The introduction of prosthetic biomaterials revolutionized hernia surgery with the concept of a tension-free repair. The subsequent rate of recurrence has been lowered to less than 10%. However, the required dissection of wide areas of soft tissue for mesh placement contribute to an incidence of wound infections and wound-related complications of 12% or greater. These problems were part of the impetus to develop minimally invasive techniques for ventral herniorrhaphy.

The laparoscopic repair of ventral hernias is rapidly evolving with patient and surgeon interest in less morbid herniorrhaphies and the appeal of minimally invasive surgery. The technique is based on the open, preperitoneal repair described by Rives and Stoppa. The placement of a large mesh in the preperitoneal location allows for an even distribution of forces along the surface area of the mesh, which may account for the strength of the repair and the decreased recurrence rates associated with it. The minimally invasive approach embraces the concept that a retromuscular mesh repair may be more durable, although the mesh is placed one layer deeper on an intact peritoneum in comparison to the open technique. The technique incorporates other fundamental components of the open repair such as wide mesh overlap of the defect and the use of transabdominal fixation sutures and spiral tacks to secure the mesh.

While the laparoscopic approach to ventral hernia repair has been documented as safe and effective, with low recurrence rates and minimal patient morbidity, some patients complain of significant post-operative pain for up to 1-3 months after surgery. The exact cause of this postoperative discomfort has not been clearly elucidated. Several hypotheses exist. Some feel that the extensive adhesiolysis required for incisional hernia repair causes significant peritoneal irritation that is exacerbated with the placement of intraperitoneal mesh. Others implicate the spiral tacks placed through the mesh into the peritoneum as sources of persistent discomfort. While others feel that the transabdominal fixation sutures are the localizing site for the accompanying postoperative pain. Transabdominal suture site pain after laparoscopic ventral hernia repair is not uncommon, and occurred in 23% of patients in one series.8 The transabdominal fixation suture sites are those incisions where sutures are placed to secure the mesh placed during laparoscopic ventral hernia repair to the anterior abdominal wall. The sutures are placed in a "clockwise" manner approximately every 4 to 5 cm at the periphery of the mesh as well as 5 mm spiral tacks to hold it in place until fibrocollagenous ingrowth secures the mesh to the abdominal wall. This persistent abdominal pain has been documented as a minor long-term complication resulting from laparoscopic ventral hernia repair, but it can be troublesome for patients in the immediate postoperative period.

The most effective method for managing this postoperative pain has not been defined.

The goal of postoperative care is to minimize the amount of pain a patient experiences following surgery and to help the patient make a quick recovery that leads to a shorter hospital stay free of complications and an earlier return to self-reliance. The most common treatment for pain after operation is opioid analgesic drug administration. Opioids are associated with undesirable side effects such as respiratory depression, nausea and vomiting, itching, increased duration of postoperative ileus, and delay in discharge. These side effects can be decreased with a reduction in the amount of opioid drugs utilized. Additionally, systemic narcotics may not optimize pain management in a specific region of the body because of its centralized effect. This may lead to a decreased mentation, reduced mobility, and a slower return to normal activities. Because a reduction of the daily consumption of narcotics is often associated with a decrease in analgesia, many other treatments for postoperative pain have been evaluated. For example, epidural analgesia is effective but the catheter needs to be placed preoperatively, is fairly invasive method, and the maintenance of the epidural treatment can be time consuming and expensive. Many studies have found clinical pain management benefits to the use of local analgesia, as measured by the use of less post-operative pain medication and more favorable ratings on pain intensity scales. Recently, a new method of delivering continuous wound infiltration with a solution of local anesthetic through an indwelling irrigation apparatus has been used in an attempt to reduce early postoperative discomfort in patients after thoracotomy, donor nephrectomy, and open inguinal hernia repair. These prospective randomized double blind studies universally report decreased postoperative discomfort and limited usage of opioids with the usage of these novel catheters.

In this study, the goal is to minimize postoperative pain so that post-operative narcotic requirements will be unnecessary or required less frequently. The infusion of a local anesthetic immediately following the surgical procedure is intended to allow the body tissues to react more favorably to surgical stress and reduce early postoperative pain.

The primary hypothesis is that continuous infusion of a local anesthetic along the edges of the mesh near the transabdominal fixation sutures and spiral tacks placed to secure mesh to the anterior abdominal wall will both subjectively and objectively improve postoperative pain control following laparoscopic ventral hernia repair. A secondary hypothesis is that pulmonary function and bowel function postoperatively will recover faster with the use of a continuous infusion of local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic ventral hernia repair
* Consent obtained

Exclusion Criteria:

* Under 18 years
* Allergic to Bupivacaine
* significant liver or renal disease
* Contraindication to PCA
* Current daily opioid usage
* History of substance abuse disorders
* Dx of chronic pain syndrome
* Daily usage of NSAIDs or COX 2 inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Place an elastomeric infusion catheter superficial to the mesh at the conclusion of the laparoscopic ventral hernia repair and compare the following to a group that receives a placebo infusion of saline: | 3 months
Measuring: Visual Analog Pain Scale, Short-Form McGill Pain Questionnaire, Present Pain Intensity, Quantity of narcotic consumption | 3 months

SECONDARY OUTCOMES:
Assess differences in postoperative pulmonary mechanics between the treated and nontreated groups by measuring the changes in maximal inspiratory volumes from baseline. | 3 months
The return of bowel function: Day of Flatus, Tolerating Regular Diet, Length of hospital stay | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Rosen, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States